CLINICAL TRIAL: NCT01734330
Title: Efficacy of Cognitive Behaviour Therapy Associated to Nicotine Replacement in Tobacco Cessation: a Randomised Open Label Clinical Trial
Brief Title: Cognitive Behaviour Therapy and Nicotine Replacement to Increase Tobacco Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 119/2010
Record Dates: First submitted 2012-11-22; First posted 2012-11-27 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Smokers
Keywords: behavior cognitive therapy; Smokers; randomized clinical trial
MeSH Terms: interventions — Cognitive Behavioral Therapy; Population Groups; Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive behavior therapy (Experimental): Cognitive behavior therapy for 6 weeks associated to nicotine replacement for 12 weeks
  Interventions: Behavioral: Cognitive behavioral therapy in group; Drug: Nicotine replacement
- Nicotine replacement (Other): Nicotine replacement for 12 weeks
  Interventions: Drug: Nicotine replacement

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy in group
  Arms: Cognitive behavior therapy
Drug: Nicotine replacement

SUMMARY:
Background: Pharmacological strategies to improve smoking cessation have been largely studied. The efficacy of cognitive behavior therapy associated to nicotine replacement in tobacco cessation has not yet been demonstrated.

Objective: Evaluate if cognitive behavior therapy during six weeks associated to nicotine replacement for twelve weeks is able to contribute to tobacco cessation at the end of 52 weeks.

Methods: Multicentre, open-label, and pragmatic randomized controlled trial will include 334 patients. Analysis will follow intention-to-treat principle.

Patients older than 18 years old and who had smoked at least 5 cigarettes in the past year before randomization will be included.

All of them will receive nicotine replacement therapy with patches and gum. They will be randomized 1:1 ratio to attend or not cognitive behavior therapy once a week for the first six weeks of the treatment. Every two weeks all of the patients will be evaluated by a physician in order to access any adverse effects from the nicotine replacement.

All patients will have carbon monoxide levels accessed at baseline and after 6 weeks. Telephonic interview will be done at 16, 28, and 52 weeks to access the rates of tobacco cessation, relapses episodes and abstinence maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Smokers (≥ 5 cigarettes/day during the previous year) who had not had a period of abstinence greater than 3 months before randomization
* Age ≥ 18 years < 75 years;
* Capable of reading and understanding Portuguese;
* Willing to quit smoking.

Exclusion Criteria:

* Dementia;
* Alcoholism;
* Regular use of illicit drugs;
* Panic disorders;
* Psychosis;
* Current pregnancy;
* History of bipolar disturbance;
* Contraindication to nicotine patches;
* Prior use of bupropion and/or varenicline in the previous 12 months before randomization;
* Patients who refused to provide informed consent;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-07; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Smoking cessation | 52 weeks

SECONDARY OUTCOMES:
Levels of anxiety | 6 weeks
  Evaluated by the State-Trait Anxiety Inventory
Levels of depression | 6 weeks
  Evaluated by Beck Depression Inventory
Smoking Relapse rates | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ismael, Study Chair — Hospital do Coração
Locations (2):
- Brazil (2):
  - Instituto de Medicina Integral Professor Fernando Figueira - IMIP, Recife, Pernanbuco
  - Hospital do Coração, São Paulo, São Paulo